CLINICAL TRIAL: NCT01146600
Title: Clarithromycin for the Treatment of Hypersomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lynn Marie Trotti (Other)
Responsible Party: Sponsor-Investigator, Lynn Marie Trotti, Assistant Professor of Neurology, Emory University
Organization: Emory University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00044170
Record Dates: First submitted 2010-06-15; First posted 2010-06-17 (Estimated); Results first posted 2014-06-12 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Hypersomnia; Idiopathic Hypersomnia; Narcolepsy
Keywords: Primary hypersomnia; CNS hypersomnia; hypersomnia; idiopathic hypersomnia; clarithromycin; Narcolepsy without Cataplexy
MeSH Terms: conditions — Disorders of Excessive Somnolence; Idiopathic Hypersomnia; Narcolepsy | interventions — Clarithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Random Group A (Experimental): Subjects will be randomized to group A or group B. The order of presentation of placebo and clarithromycin will be opposite in these two groups, but investigators and subjects will remain blinded to group allocation and order of treatment presentation within the groups.
  Interventions: Drug: Clarithromycin followed by placebo
- Random Group B (Experimental): Subjects will be randomized to group A or group B. The order of presentation of placebo and clarithromycin will be opposite in these two groups, but investigators and subjects will remain blinded to group allocation and order of treatment presentation within the groups.
  Interventions: Drug: Placebo then Clarithromycin

INTERVENTIONS:
Drug: Clarithromycin followed by placebo — Clarithromycin 500 mg po bid for two weeks, then one week with no medication, then matched placebo po bid for two weeks.
  Other Names: Biaxin
  Arms: Random Group A
Drug: Placebo then Clarithromycin — Matched placebo po bid for two weeks, then one week with no intervention, then clarithromycin 500 mg po bid for two weeks
  Other Names: Biaxin
  Arms: Random Group B

SUMMARY:
The term 'hypersomnia' describes a group of symptoms that includes severe daytime sleepiness and sleeping long periods of time (more than 10 hours per night). Sometimes, hypersomnia is caused by a problem with the quality of sleep occurring at night, for instance when nighttime sleep is disrupted by frequent breathing pauses. In other cases, however, hypersomnia occurs even when nighttime sleep is of good quality. These cases of hypersomnia are presumed to be a symptom of brain dysfunction, and so are referred to as hypersomnias of central (i.e., brain) origin.

The causes of most of these central hypersomnias are not known. However, our group has recently identified a problem with the major brain chemical responsible for sedation, known as GABA. In a subset of our hypersomnia patients, there is a naturally-occurring substance that causes the GABA receptor to be hyperactive. In essence, it is as though these patients are chronically medicated with Valium (or Xanax or alcohol, all substances that act through the GABA system), even though they do not take these medications.

Current treatment of central hypersomnias is limited. For the fraction of cases with narcolepsy, there are FDA-approved, available treatments. However, for the remainder of patients, there are no treatments approved by the FDA. They are usually treated with medications approved for narcolepsy, but sleep experts agree that these medications are often not effective for this group of patients.

Based on our understanding of the GABA abnormality in these patients, we evaluated whether clarithromycin (an antibiotic approved by the FDA for the treatment of infections) would reverse the GABA abnormality. In a test tube model of this disease, clarithromycin does in fact return the function of the GABA system to normal. The investigators have treated a few patients with clarithromycin and most have felt that their hypersomnia symptoms improved with this treatment.

To determine whether clarithromycin is truly beneficial for central hypersomnia, this study will compare clarithromycin to an inactive pill (the placebo). All subjects will receive both clarithromycin and the placebo at different times, and their reaction times and symptoms will be compared on these two treatments to determine if one is superior. If this study shows that clarithromycin is more effective than placebo in the treatment of hypersomnia, it will identify a potential new therapy for this difficult-to-treat disorder.

DETAILED DESCRIPTION:
Central hypersomnias are characterized by severe excessive daytime sleepiness despite long sleep periods (>10 hours/night) and the absence of nocturnal sleep pathology. They preferentially affect young adults, may result in loss of employment, and can lead to motor vehicle accidents (1). Despite these health, safety, and quality of life consequences, there are no FDA-approved therapies for several forms of central hypersomnia, including idiopathic hypersomnia (IH). Currently, IH is treated using therapies approved for narcolepsy, despite a lack of clinical trial data and a consensus that treatment response is poor (2). Treatments include traditional psychostimulants (e.g., amphetamine derivatives) as well as wake-promoting agents with unknown mechanisms of action such as modafinil and sodium oxybate. In addition to side effects including high abuse potential, tachycardia, and altered mental status, treatments are often ineffective and substantial residual sleepiness frequently persists despite poly-therapy.

The investigators hypothesize that pathology in the GABA neurotransmitter system, the brain's major inhibitory system, underlies these central hypersomnias. Currently, there are no hypersomnia therapies that are GABA-antagonists. However, the macrolide antibiotic clarithromycin has been shown to have GABA-modulating properties, resulting in the development of insomnia or mania in a subset of patients. Clarithromycin is therefore a potentially viable, promising therapeutic agent for hypersomnia related to positive modulation of the GABAA receptor. Open-label use of clarithromycin in six hypersomnia patients with known (n = 4) or suspected (n = 2) excess GABAA potentiation resulted in marked improvements in vigilance, as measured on the psychomotor vigilance task (PVT) (unpublished data). The investigators therefore propose a pilot, crossover trial comparing clarithromycin to placebo for the treatment of hypersomnia in patients with excess GABAA potentiation. The primary endpoint will be a decrease in PVT reaction time. Secondary endpoints will include a decrease in PVT lapses and changes in Epworth, Stanford, and FOSQ sleep scales. Successful results from this trial would provide early evidence for a more rational and efficacious treatment for hypersomnia that could avoid the potential abuse, toxicities, and treatment failures associated with traditional treatments.

This will be a pilot crossover trial of clarithromycin and placebo to treat central hypersomnia. Subjects who are untreated for hypersomnia or who experience persistent symptoms despite traditional therapies will be eligible. Subjects who are on medication for hypersomnia at the beginning of the study will be asked to maintain stable doses of these medications for one month before and throughout the study period. Twenty subjects will be assessed at baseline and one and two weeks after being on each study drug (clarithromycin 500 mg bid and matched placebo bid). After two weeks on study drug, they will undergo a one week washout period, then change to the other study drug for an additional two weeks. Patients will be randomized to order of presentation of study drugs such that ten subjects will be randomized to each group. Random sequence generation will be performed our pharmacy. All study investigators and subjects will remain blinded to group assignment.

ELIGIBILITY:
Inclusion Criteria:

* Hypersomnia (meeting clinical criteria for Idiopathic hypersomnia with or without long sleep time, narcolepsy lacking cataplexy, or symptomatic hypersomnia not meeting ICSD criteria)
* evidence for GABA-related abnormality, as demonstrated by in-house, in vitro assay
* age > 18
* high performance liquid chromatography/liquid chromatography tandem mass spectrometry verification of the absence of exogenous benzodiazepines

Exclusion Criteria:

* Contraindications to use of clarithromycin (pregnancy, severe renal impairment, history of QT prolongation, hypomagnesemia, hypokalemia, bradycardia, history of myocardial infarction or cardiomyopathy, myasthenia gravis, age > 70)
* Current use of cisapride, pimozide, astemizole, terfenadine, colchicines, and ergotamine or dihydroergotamine
* Current use of benzodiazepines or benzodiazepine-receptor agonists
* moderate or severe sleep apnea (RDI > 15/hr), severe periodic limb movement disorder (PLMI > 30/hr)
* diagnosis of narcolepsy with cataplexy, as determined by cerebrospinal hypocretin levels
* metabolic disorders such as anemia, severe iron deficiency, B12 deficiency, or hypothyroidism that may explain symptoms of hypersomnia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Marie Trotti, MD, Principal Investigator — Emory University
Locations (1):
- Emory Sleep Center, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Trotti LM, Becker LA, Friederich Murray C, Hoque R. Medications for daytime sleepiness in individuals with idiopathic hypersomnia. Cochrane Database Syst Rev. 2021 May 25;5(5):CD012714. doi: 10.1002/14651858.CD012714.pub2. PMID 34031871
- [Derived] Trotti LM, Saini P, Bliwise DL, Freeman AA, Jenkins A, Rye DB. Clarithromycin in gamma-aminobutyric acid-Related hypersomnolence: A randomized, crossover trial. Ann Neurol. 2015 Sep;78(3):454-65. doi: 10.1002/ana.24459. Epub 2015 Jun 30. PMID 26094838

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Most subjects were recruited from the patient population of a single Sleep Center affiliated with Emory University School of Medicine. One subject contacted investigators for participation after reading of the study on clinicaltrials.gov. The first patient was recruited 3/5/11 and the final patient completed the study on 9/28/12.
Pre-assignment Details: All subjects underwent screening laboratories after enrollment but before beginning medication. In the case of abnormal laboratory results (n = 2), subjects did not begin treatment with either study drug (clarithromycin or placebo). One patient dropped out after consent but before randomization (because of scheduling conflict).
Groups:
- Clarithromycin, Then Placebo: Subjects randomized to receive clarithromycin first (for two weeks), then matched placebo (for an additional two weeks, following the washout)
- Placebo, Then Clarithromycin: Subjects randomized to receive placebo first (for two weeks), then clarithromycin (for an additional two weeks, following the washout)
Period: Period 1 (Weeks 1 & 2)
Arm/Group | Clarithromycin, Then Placebo | Placebo, Then Clarithromycin
Started | 13 | 10
Completed | 10 | 10
Not Completed | 3 | 0
Period: Washout (Week 3)
Arm/Group | Clarithromycin, Then Placebo | Placebo, Then Clarithromycin
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Period 2 (Weeks 4 & 5)
Arm/Group | Clarithromycin, Then Placebo | Placebo, Then Clarithromycin
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Clarithromycin, Then Placebo: Subjects will be randomized to group A or group B. The order of presentation of placebo and clarithromycin will be opposite in these two groups, but investigators and subjects will remain blinded to group allocation and order of treatment presentation within the groups.
  Clarithromycin followed by placebo : Clarithromycin 500 mg po bid (with breakfast and lunch) for two weeks, then one week with no medication, then matched placebo po bid (with breakfast and lunch) for two weeks.
- Placebo, Then Clarithromycin: Subjects will be randomized to group A or group B. The order of presentation of placebo and clarithromycin will be opposite in these two groups, but investigators and subjects will remain blinded to group allocation and order of treatment presentation within the groups.
  Placebo then Clarithromycin : Matched placebo po bid (with breakfast and lunch) for two weeks, then one week with no intervention, then clarithromycin 500 mg po bid (with breakfast and lunch) for two weeks
- Total: Total of all reporting groups
Arm/Group | Clarithromycin, Then Placebo | Placebo, Then Clarithromycin | Total
Number analyzed (Participants) | 13 | 10 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 10 | 23
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (13.4) | 34.7 (14.5) | 34.2 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 13 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Psychomotor Vigilance Task (PVT) Reaction Time
Description: Median reaction time on the PVT at the end of the second week of treatment. Lower values reflect faster reaction times (I.e., greater vigilance).
  Note that the PVT provides a median of reaction times to all stimuli (~100) presented during the 10 minute PVT test. Each subject had two PVT tests at each visit, resulting in two median values. These were averaged, and then, for the purposes of this outcome, we then obtained the MEAN across multiple subjects for each condition (baseline, clarithromycin week 2, placebo week 2)
Time Frame: week 2 of each intervention
Population: Analysis was performed on all subjects who took both study drugs (i.e., clarithromycin and placebo)
Measure: Mean (Standard Deviation); unit: Msec
Groups:
- Clarithromycin: Clarithromycin 500 mg with breakfast and 500 mg with lunch for two weeks
- Placebo: Matched placebo with breakfast and with lunch for two weeks
- Baseline: Baseline values (prior to first study drug) for the 20 subjects who completed both treatment arms.
Arm/Group | Clarithromycin | Placebo | Baseline
Number analyzed (Participants) | 20 | 20 | 20
Msec | 279.1 (77.3) | 311.6 (114.1) | 333.8 (291.4)
Statistical Analysis 1: Comparison: Clarithromycin vs Placebo vs Baseline; Test type: Superiority or Other; p = 0.47, ANOVA; ANOVA, comparing baseline, clarithromycin, and placebo

2. Secondary Outcome: PVT Median Reaction Time at Week 1
Description: median reaction time on the PVT at week 1 of each intervention. Lower values reflect faster reaction times (i.e., better vigilance)
  Note that the PVT provides a median of reaction times to all stimuli (~100) presented during the 10 minute PVT test. Each subject had two PVT tests at each visit, resulting in two median values. These were averaged, and then, for the purposes of this outcome, we then obtained the MEAN across multiple subjects for each condition (baseline, clarithromycin week 1, placebo week 1)
Time Frame: week 1
Population: Analysis was performed on all subjects who took both study drugs (i.e., clarithromycin and placebo)
Measure: Mean (Standard Deviation); unit: Msec
Arm/Group | Clarithromycin | Placebo | Baseline
Number analyzed (Participants) | 20 | 20 | 20
Msec | 285.4 (71.3) | 308.4 (120.6) | 333.8 (291.4)
Statistical Analysis 1: Comparison: Clarithromycin vs Placebo vs Baseline; Test type: Superiority or Other; p = 0.63, ANOVA; ANOVA comparing baseline, clarithromycin, and placebo

3. Secondary Outcome: PVT Number of Lapses
Description: Number of lapses (no response for > 500 msec) on the PVT, averaged by subject across all administrations for a given drug condition (i.e. administered twice at baseline, four times on clarithromycin (twice during week 1 and twice during week 2), and four times on placebo (twice during week 1 and twice during week 2)). Higher numbers indicate worse vigilance.
Time Frame: baseline, then after 1 week and 2 weeks on each study drug
Population: Analysis was performed on all subjects who took both study drugs (i.e., clarithromycin and placebo)
Measure: Mean (Standard Deviation); unit: Number of lapses
Arm/Group | Clarithromycin | Placebo | Baseline
Number analyzed (Participants) | 20 | 20 | 20
Number of lapses | 5.7 (11.3) | 10.3 (18.7) | 6.5 (16.9)
Statistical Analysis 1: Comparison: Clarithromycin vs Placebo vs Baseline; Test type: Superiority or Other; p = 0.64, ANOVA; ANOVA comparing baseline, clarithromycin, and placebo

4. Secondary Outcome: Epworth Sleepiness Scale
Description: Scores on the Epworth Sleepiness Scale (ESS) were averaged by subject across all administrations for a given drug condition (i.e. administered twice on clarithromycin (once during week 1 and once during week 2) and twice on placebo (once during week 1 and once during week 2)).
  ESS scores can range from 0 to 24. Higher scores indicate higher levels of sleepiness.
Time Frame: baseline, then after 1 week and 2 weeks on each study drug
Population: Analysis was performed on all subjects who took both study drugs (i.e., clarithromycin and placebo)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clarithromycin | Placebo | Baseline
Number analyzed (Participants) | 20 | 20 | 20
units on a scale | 10.1 (5.4) | 14.1 (3.7) | 15.0 (2.3)
Statistical Analysis 1: Comparison: Clarithromycin vs Placebo vs Baseline; Test type: Superiority or Other; p = 0.002, ANOVA; ANOVA comparing baseline, clarithromycin, and placebo

5. Secondary Outcome: FOSQ
Description: Scores on the Functional Outcomes of Sleep Questionnaire (FOSQ) were averaged by subject across all administrations for a given drug condition (i.e. administered twice on clarithromycin (once during week 1 and once during week 2) and twice on placebo (once during week 1 and once during week 2)).
  Scores on the FOSQ can range from 5 to 20. Higher FOSQ scores indicate less impairment due to sleepiness.
Time Frame: baseline, then after 1 week and 2 weeks on each study drug
Population: Analysis was performed on all subjects who took both study drugs (i.e., clarithromycin and placebo)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clarithromycin | Placebo | Baseline
Number analyzed (Participants) | 20 | 20 | 20
units on a scale | 16.6 (2.4) | 14.4 (2.7) | 13.9 (2.0)
Statistical Analysis 1: Comparison: Clarithromycin vs Placebo vs Baseline; Test type: Superiority or Other; p = 0.002, ANOVA; ANOVA comparing baseline, clarithromycin, and placebo

6. Secondary Outcome: SF-36, Vitality Subscale
Description: The SF-36 is a health outcome scale with multiple subsections. Subjects were administered the entire SF-36; this analysis is of the vitality subscore provided by this scale. Scores were averaged by subject across all administrations for a given drug condition (i.e. administered once at baseline, twice on clarithromycin (once during week 1 and once during week 2) and twice on placebo (once during week 1 and once during week 2)).
  The vitality subscore is calculated using four questions from the SF-36, and can range from 0 to 100. Higher scores reflect more vitality.
Time Frame: baseline, then after 1 week and 2 weeks on each study drug
Population: Analysis was performed on all subjects who took both study drugs (i.e., clarithromycin and placebo)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clarithromycin | Placebo | Baseline
Number analyzed (Participants) | 20 | 20 | 20
units on a scale | 48.9 (26.9) | 28.0 (22.5) | 25.0 (21.6)
Statistical Analysis 1: Comparison: Clarithromycin vs Placebo vs Baseline; Test type: Superiority or Other; p = 0.01, ANOVA; ANOVA comparing baseline, clarithromycin, and placebo

7. Secondary Outcome: PSQI
Description: Scores on the Pittsburgh Sleep Quality Index (PSQI), a questionnaire based assessment of sleep quality. Scores were averaged by subject across all administrations for a given drug condition (i.e. administered twice on clarithromycin (once during week 1 and once during week 2) and twice on placebo (once during week 1 and once during week 2)).
  Scores on the PSQI can range from 0 to 21. Higher scores indicate poorer sleep quality.
Time Frame: baseline, then after 1 week and 2 weeks on each study drug
Population: Analysis was performed on all subjects who took both study drugs (i.e., clarithromycin and placebo)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clarithromycin | Placebo | Baseline
Number analyzed (Participants) | 20 | 20 | 20
units on a scale | 5.8 (3.9) | 6.3 (2.8) | 6.7 (3.5)
Statistical Analysis 1: Comparison: Clarithromycin vs Placebo vs Baseline; Test type: Superiority or Other; p = 0.76, ANOVA; ANOVA comparing baseline, clarithromycin, and placebo

ADVERSE EVENTS:
Arm/Group | Clarithromycin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 21/22 | 15/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Clarithromycin (N=22) | Placebo (N=20)
abdominal pain (Gastrointestinal disorders) | 3 | 1
anxiety (Psychiatric disorders) | 1 | 1
bad taste or smell (General disorders) | 15 | 0
bloating/gas (Gastrointestinal disorders) | 2 | 1
chest discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
diarrhea (Gastrointestinal disorders) | 4 | 5
dizziness (Nervous system disorders) | 1 | 1
feeling "jittery" or "hyper" (Nervous system disorders) | 3 | 1
headache (Nervous system disorders) | 3 | 5
hiccups (General disorders) | 0 | 1
change in appetite (increase or decrease) (Gastrointestinal disorders) | 2 | 1
sweating, flushing, or feeling hot (General disorders) | 2 | 1
insomnia (Nervous system disorders) | 6 | 3
knee pain (Musculoskeletal and connective tissue disorders) | 0 | 1
nausea (Gastrointestinal disorders) | 7 | 3
nose bleed (General disorders) | 2 | 0
symptoms of upper respiratory infection (Infections and infestations) | 0 | 3
syncope (Cardiac disorders) | 0 | 1
tremor (Nervous system disorders) | 1 | 1
unspecified gastrointestinal distress (Gastrointestinal disorders) | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes